CLINICAL TRIAL: NCT00978484
Title: A Head-to-head Comparison of Virtual Reality Treatment for Post Traumatic Stress Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Defense Centers of Excellence for Psychological Health and Traumatic Brain Injury (U.S. Federal Agency); The Geneva Foundation (Other); Marine Corps Base Camp Pendleton (Other); Naval Hospital Camp Pendleton (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert McLay, PI, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-08-1-0755; W81XWH-08-1-0755
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Depression; Anxiety; Virtual Reality; Computer Therapy; Exposure Therapy; Prolonged Exposure; Military Medicine; Combat; Iraq; Afghanistan; Air Force Personnel; Armed Forces Personnel; Army Personnel; Coast Guard; psychology; military psychiatry; combat disorders; combat neurosis; Marines; Military; Navy Personnel; Sailors; Soldiers
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Combat Disorders | interventions — beta-Aminoethyl Isothiourea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Static Virtual Reality (Active Comparator): Exposure Therapy using a still computer image
  Interventions: Behavioral: Augmented Exposure Therapy
- Dynamic Virtual Reality (Experimental): Virtual Reality Exposure Therapy using full, immersive Virtual Reality
  Interventions: Behavioral: Virtual Reality Exposure Therapy - Dynamic

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy - Dynamic — 10 weeks of Virtual Reality Exposure using full, immersive VR
  Other Names: VRE; VRET
  Arms: Dynamic Virtual Reality
Behavioral: Augmented Exposure Therapy — Exposure Therapy augmented with a still computer image
  Other Names: AET; Static VRE; Prolonged Exposure; PE
  Arms: Static Virtual Reality

SUMMARY:
Therapy that uses Virtual Reality (VR) has been shown to help in the treatment of Post Traumatic Stress Disorder (PTSD). It is unclear what role the VR simulator itself plays in recovery. This study is examining if full-immersion in VR causes greater improvement in PTSD symptoms than does similar therapy that uses a simple, static, computer image.

DETAILED DESCRIPTION:
Exposure Therapy (ET) is the current gold standard for treating Post Traumatic Stress Disorder (PTSD). Although ET has the best evidence in its favor, it is also clear that the treatment is less than perfect in achieving remission of PTSD. Attempts have been made to improve on traditional ET by augmenting the exposure using Virtual Reality (VR). Open label trials of VR assisted ET (VRET) showed this method to be safe and effective, and suggested remission rates that were higher than normally seen with ET alone. For the treatment of phobias, head to head comparison with traditional ET has shown VRET to be superior. For PTSD, trials that directly pit VRET against traditional ET, and against other traditional therapy, are ongoing, but it is already clear that some individuals who fail to respond to traditional ET do get better once VR is added. Lost in the rush to develop VRET, however, has been any direct testing of its signature aspect, the VR itself. There are theoretical reasons to believe that VR might enhance ET in special ways. However there are other reasons to believe that any form of Augmented Exposure Therapy (AET) that introduced sights and sounds from the trauma would do just as well. VR, although exciting, is expensive, cumbersome, and not available at most treatment facilities. If similar effects could be achieved using more primitive technology, it would open up the possibility of enhanced ET to a much wider range of patients. Conversely, if VRET were shown to be superior to simplified AET, it would argue for a unique role of VR in psychotherapy. Not only would this be theoretically important for neuroscientists, it would indicate VRET as a "platinum" standard for treating PTSD. For the past four years, programs at Naval Medical Center San Diego (NMCSD) and Naval Hospital Camp Pendleton have collaborated with VR companies and researcher to build and test VR systems to treat PTSD in Service Members returning from Iraq and Afghanistan. NMCSD thus has the experience to perform the necessary experiments. The existing equipment also means that NMCSD has the unique ability to carry out such a test without any additional input from the companies that make VR systems. We propose to perform a randomized, head-to-head study that compares VRET to AET. We propose to perform a randomized, head-to-head study that compares VRET to AET. Up to 300 patients would be recruited with the goal of treating 40 patients with VR and 40 patients with the control (AET) therapy. The same techniques, measures, and controls would be used that NMCSD has already put in place to develop VRET for PTSD. Also, a cost-benefit analysis would be used to determine the benefits of VRET.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be eligible to receive care at NMCSD or Camp Pendleton, willing and able to give informed consent, aged 18 to 60, have a PTSD diagnosis from combat operations in Iraq or Afghanistan based on DSM-IV criteria and Clinician Administered PTSD Scale (CAPS) score greater than 40, have an index trauma that occurred in Iraq or Afghanistan, be medically able to tolerate exposure treatment and physically able to don virtual reality headset and physiological monitoring equipment as assed by their medical provider, be willing and able to give up alcohol and/or other intoxicating substances within 12 hours of a VR treatment session, and be able to see, hear, and smell

Exclusion Criteria:

Subjects would be excluded or dropped from the study if they exhibit psychosis, mania, epilepsy, have current suicidal intent, are less than 30 days from a psychiatric hospitalization or suicide attempt, meet criteria for current, active substance dependence, use an intoxicating substance within 12 hours of a treatment session, or have another condition or event that the treating provider or medical monitor consider to be a safety hazard within the study. Subjects may also drop out of the study at any point with the assurance that they will be referred to other care as needed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PSTD Scale (CAPS) | Post Tx, and 3 month follow up

SECONDARY OUTCOMES:
PTSD Checklist, Military Version (PCL-M): | Post Tx, and 3 month follow up
The Patient Health Questionnaire 9 (PHQ-9): | same
Beck Anxiety Inventory (BAI): | same
Behavioral Reactivity Test (BRT) | same
Automated Neuropsychological Assessment Metric (ANAM) | same
Mini International Neuropsychiatric Interview (MINI) | same
Shehan Disability Scale (SDS) | same

CONTACTS AND LOCATIONS:
Overall Officials: Robert N McLay, MD/PhD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (2):
- United States (2):
  - Camp Pendlton, Camp Pendlton, California
  - Naval Medical Center San Diego (NMCSD), San Diego, California